CLINICAL TRIAL: NCT06850844
Title: Impact of Recruitment Maneuvers and PEEP-guided Electrical Impedance Tomography on Regional Ventilation, Gas Exchange, and Pulmonary Mechanics in in Abdominal Laparoscopic Surgery Patients
Brief Title: Recruitment Maneuvers and PEEP-guided Electrical Impedance Tomography for Abdominal Laparoscopic Surgery Patients
Acronym: PEEP-EIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nguyen Dang Thu (Other)
Collaborators: Bach Mai Hospital (Other); Hanoi Medical University (Other)
Responsible Party: Sponsor-Investigator, Nguyen Dang Thu, Ph.D; M.D., Vietnam Military Medical University
Organization: Vietnam Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HuyenGMHS 5509/BM-HDDD; No.5509/BM-HDDD (Other: Bach Mai Hospital)
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Surgery; Positive End-Expiratory Pressure; Electrical Impedance Tomography
Keywords: Laparoscopic Surgery; Positive End-Expiratory Pressure; Recruitment Maneuver; electrical impedance tomography; blood oxygenation; regional ventilation; pulmonary mechanics

STUDY DESIGN:
Intervention Model Description: Prospective, single center, randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Patients were applied recruitment maneuvers and EIT-guided PEEP during ventilation during general anesthesia.
  Interventions: Device: electrical impedance tomography
- Control Group (Placebo Comparator): Patients will receive a constant PEEP of 5 cm H2O without RMs throughout the entire intraoperative ventilation period
  Interventions: Device: Conventional Ventilation

INTERVENTIONS:
Device: electrical impedance tomography — The individualized high PEEP with RMs group commences with a PEEP of 5 cm H2O and undergo an RM followed by a decremental PEEP trial. Pressure-controlled ventilation mode is set with a respiratory rate of 16 breaths per minute and ΔP=15 (ΔP is calculated by subtracting PEEP from the plateau pressure (Pplat). In intervals of 5 breaths, PEEP is incrementally increased by 5 cm H2O, starting at 5 cm H2O and reaching up to 20 cm H2O. The decremental PEEP trial is immediately performed following the first RM, beginning at a PEEP of 20 cm H2O with a respiratory rate of 15 breaths per minute. Every 30 seconds, PEEP is decreased by increments of 2 cm H2O until it reaches a minimum of 6 cm H2O. This decremental PEEP trial is succeeded by a second RM, after which the individualized PEEP level will be established as determined by the decremental PEEP trial and sustained until the completion of ventilation.
  Arms: Intervention Group
Device: Conventional Ventilation — Ventilation is set in volume-controlled mode with a tidal volume of 7 ml/kg predicted body weight (PBW), the respiratory rate is adjusted to target normocapnia (end-tidal carbon dioxide partial pressure between 35 and 45 mmH), an inspiratory to expiratory ratio of 1:2, and a PEEP of 5 cmH2O.
  Arms: Control Group

SUMMARY:
Abdominal laparoscopy is widely utilized due to its benefits, including minimal invasiveness, improved cosmetic outcomes, and shorter hospital stays. However, the use of intraoperative pneumoperitoneum and general anesthesia with mechanical ventilation may lead to postoperative pulmonary complications, such as atelectasis. This condition can result in diminished respiratory mechanics and impaired gas exchange.

In recent years, intraoperative lung-protective mechanical ventilation techniques, including recruitment maneuvers (RMs) and positive end-expiratory pressure (PEEP) strategies, have gained popularity. These approaches aim to prevent the repeated collapse and reopening of alveoli, thereby reducing the risk of atelectasis. Nonetheless, determining the optimal PEEP level for individual patients remains a complicated and unresolved issue.

Electrical impedance tomography (EIT) is a bedside imaging technique that assesses regional ventilation distribution, providing a method for personalizing PEEP settings in mechanically ventilated patients. By addressing the competing risks of alveolar overdistension and collapse, EIT enhances the precision of PEEP titration.

This study aims to compare the effects of recruitment maneuvers and EIT-guided PEEP selection against conventional ventilation on regional ventilation, gas exchange, and pulmonary mechanics in patients undergoing abdominal laparoscopic surgery.

DETAILED DESCRIPTION:
This is a prospective, single-center, randomized controlled trial designed to evaluate the effects of recruitment maneuvers and EIT-guided PEEP selection against conventional ventilation on regional ventilation, gas exchange, and pulmonary mechanics in patients undergoing abdominal laparoscopic surgery. Adult patients undergoing abdominal laparoscopic surgery will be enrolled in the study. Patients in the intervention group will receive intraoperative regular recruitment maneuvers and PEEP titrated using EIT with a stepwise decremental PEEP trial, while those in the control group will have a constant PEEP of 5 cmH2O. The primary outcomes are regional ventilation, blood oxygenation, and pulmonary mechanics. Secondary outcomes include hemodynamic effects, pneumothorax or barotrauma events during the intraoperative period, pulmonary complications during the first 5 days postoperative, and length of hospital stay.

Standard Ventilation Management:

Patients in both groups receive volume-controlled ventilation at the lowest possible inspired oxygen fraction (FiO2), with a minimum of 0.4, to maintain peripheral oxygen saturation (SpO2) above 92%. The inspiratory to expiratory ratio (I:E) is set at 1:2, and the respiratory rate is adjusted to achieve normocapnia, defined as an end-tidal carbon dioxide partial pressure between 35 and 45 mmHg. Tidal volume (VT) is set at 7 ml/kg predicted body weight (PBW), calculated using the following formula: for males, 50 + 0.91 × (height in centimeters - 152.4), and for females, 45.5 + 0.91 × (height in centimeters - 152.4).

Intervention Patients were randomized into either the intervention group or the control group.

Intervention Group: The individualized high PEEP with RMs group will commence with a PEEP of 5 cm H2O and will undergo an RM followed by a decremental PEEP trial. RMs are conducted only when hemodynamic stability is confirmed by the attending anesthesiologist. For this process, the ventilator is set to pressure-controlled ventilation mode, with a respiratory rate of 16 breaths per minute and ΔP=15 (ΔP is calculated by subtracting PEEP from the plateau pressure (Pplat)). In intervals of 5 breaths, PEEP is incrementally increased by 5 cm H2O, starting at 5 cm H2O and reaching up to 20 cm H2O. The decremental PEEP trial is immediately performed following the first RM, beginning at a PEEP of 20 cm H2O with a respiratory rate of 15 breaths per minute while maintaining the ventilator in pressure-controlled ventilation mode. Every 30 seconds, PEEP is decreased by increments of 2 cm H2O until it reaches a minimum of 6 cm H2O. This decremental PEEP trial is succeeded by a second RM, after which the individualized PEEP level will be established as determined by the decremental PEEP trial and sustained until the completion of ventilation.

Control Group: Patients will receive a constant PEEP of 5 cm H2O without RMs throughout the entire intraoperative ventilation period.

Rescue strategies Desaturation (defined as SpO2 ≤ 90% or if preoperative SpO2 < 90% an absolute decrease in SpO2 > 5%) If desaturations occur and there are no airway problems, severe hemodynamic impairment or ventilator malfunction, a rescue strategy is allowed by increasing FiO2 first, eventually followed by RM and PEEP increases.

Preapproved protocol deviations

If one of the following complications occurs and does not respond to conventional therapy, PEEP can be changed, according to the judgment of the anesthesiologist in charge:

(i) After PEEP titration, a mean arterial pressure (MAP) < 65 mmHg, lasting > 1 min and not responding to fluids and/or vasoactive drugs.

(ii) New arrhythmias not responding to the treatment suggested by the Advanced Cardiac Life Support guidelines.

(iii) Need for a dosage of vasoactive drugs at the highest level tolerated, according to the decision of the anesthesiologist in charge.

(iv) Need of massive transfusion, more than five units of blood to maintain hematocrit > 21% and hemoglobin> 7 mg/dL.

(v) Surgical complication resulting in a life-threatening situation. Any deviation from the protocol, excluding those mentioned above, is classified as a protocol violation. Protocol violations are to be reported and will be discussed with the data safety monitoring board.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Scheduled for abdominal laparoscopy surgery
* At increased (i.e., intermediate or high) risk of postoperative pulmonary complications according to the "Assess Respiratory Risk in Surgical Patients in Catalonia" (ARISCAT) score (≥ 26 points)
* Signed written informed consent

Exclusion Criteria:

* Major previous lung surgery (e.g., lung resection)
* Severe chronic obstructive pulmonary disease and/or severe emphysema
* Increased intracranial pressure
* Contraindications for EIT (pacemakers, automatic external defibrillators, cases of chest trauma or recent chest surgery limiting EIT belt application)
* Presence of pneumothorax that is either undrained or newly occurred.
* Unstable hemodynamics with a mean arterial pressure < 60 mmHg and unresponsive to resuscitation measures, and/or heart rate < 60 bpm.
* Pregnancy.
* Severe neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Regional Lung Ventilation | During surgery
  Evaluation of Ventilation Distribution With Electrical Impedance Tomography
Oxygenation | During surgery, and at day 1 post-operative
  PaO2/FiO2 will be evaluated via arterial blood gas analysis
Pulmonary Mechanic | During surgery
  Static Compliance

SECONDARY OUTCOMES:
Pneumothorax or barotrauma | During surgery
  New-onset of pneumothorax and barotrauma
Hemodynamic instability | During surgery
  New-onset of Bradycardia and/or hypotension
Respiratory failure | Up to 5 days after surgery
  pO2 less than 60 mm Hg (or room air oxygen saturation less than or equal to 90%), pCO2 greater than 50 mm Hg with pH less than 7.35, and signs/symptoms of respiratory distress
Bronchospasm | Up to 5 days after surgery
  Symptoms and signs of acute bronchospasm include wheezing, prolonged expiration, reduced breath sounds
Suspected pulmonary infection | Up to 5 days after surgery
  A patient should be suspected of having pneumonia when the following signs and symptoms are present. An acute cough and one of the following: new focal chest signs; dyspnoea; tachypnoea; or fever >4 days
Pulmonary infiltrate | Up to 5 days after surgery
  New pulmonary infiltrate of at least one complete lung segment with alveolar consolidation and excluding atelectasis; and presence of chest pain, temp T >38.5°C, tachypnea, wheezing, or cough.
Pleural effusion | Up to 5 days after surgery
  New-onset of Pleural effusion

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia Center, Bach Mai Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cinnella G, Grasso S, Spadaro S, Rauseo M, Mirabella L, Salatto P, De Capraris A, Nappi L, Greco P, Dambrosio M. Effects of recruitment maneuver and positive end-expiratory pressure on respiratory mechanics and transpulmonary pressure during laparoscopic surgery. Anesthesiology. 2013 Jan;118(1):114-22. doi: 10.1097/ALN.0b013e3182746a10. PMID 23196259
- [Result] Karsten J, Luepschen H, Grossherr M, Bruch HP, Leonhardt S, Gehring H, Meier T. Effect of PEEP on regional ventilation during laparoscopic surgery monitored by electrical impedance tomography. Acta Anaesthesiol Scand. 2011 Aug;55(7):878-86. doi: 10.1111/j.1399-6576.2011.02467.x. Epub 2011 Jun 9. PMID 21658014
- [Result] Nestler C, Simon P, Petroff D, Hammermuller S, Kamrath D, Wolf S, Dietrich A, Camilo LM, Beda A, Carvalho AR, Giannella-Neto A, Reske AW, Wrigge H. Individualized positive end-expiratory pressure in obese patients during general anaesthesia: a randomized controlled clinical trial using electrical impedance tomography. Br J Anaesth. 2017 Dec 1;119(6):1194-1205. doi: 10.1093/bja/aex192. PMID 29045567
- [Result] Erlandsson K, Odenstedt H, Lundin S, Stenqvist O. Positive end-expiratory pressure optimization using electric impedance tomography in morbidly obese patients during laparoscopic gastric bypass surgery. Acta Anaesthesiol Scand. 2006 Aug;50(7):833-9. doi: 10.1111/j.1399-6576.2006.01079.x. PMID 16879466